CLINICAL TRIAL: NCT04237233
Title: Intense Monitoring Study on Sintilimab Injection (Tyvyt®)
Brief Title: Intense Monitoring Study on Tyvyt
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Innovent Biologics (Suzhou) Co. Ltd. (Industry)
Responsible Party: Sponsor
Other Study IDs: CIBI308B401
Record Dates: First submitted 2019-12-31; First posted 2020-01-23 (Actual); Last update posted 2022-09-16 (Actual); Status verified 2022-09

CONDITIONS: Relapsed or Refractory Classical Hodgkin's Lymphoma
MeSH Terms: conditions — Recurrence

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The study is a multi-center, prospective, non-interventional and observational study, and will collect data on the safety and efficacy of Tyvyt® in the treatment of Chinese patients with relapsed or refractory classical Hodgkin's lymphoma.

ELIGIBILITY:
Inclusion Criteria:

Patients must be able to understand and voluntarily sign the informed consent form (ICF).

Patients must provide reliable contact information, including home phone numbers or follow-up phone number, and be voluntary to be followed up.

Patients must have agreed to use Tyvyt® to treat the target indication.

Exclusion Criteria:

Patients refuse to be included in the study or refuse to cooperate.

Patients have participated in another interventional studies within 4 weeks prior to enrollment.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The main study population is target indication patients treated with Tyvyt® within the territory of China. If any new indication is approved during the implementation of the project, and there are no special requirements for the approval, the new indication patients using Tyvyt® will also be included in the study.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2020-04-02 (Actual); Primary Completion 2023-06 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Incidence of known adverse drug reactions | During the actual Tyvyt treatment time.
Occurrence of new adverse drug reactions | During the actual Tyvyt treatment time.
Association, risk factors, severity and incidence of immune-related adverse drug reactions/events | During the actual Tyvyt treatment time.
Association, risk factors, severity and incidence of serious adverse drug reactions | During the actual Tyvyt treatment time.
Occurrence of adverse drug reactions in special population | During the actual Tyvyt treatment time.

SECONDARY OUTCOMES:
Overall survival (OS) | During the actual Tyvyt treatment time.

CONTACTS AND LOCATIONS:
Locations (1):
- Peking Union Medical College Hospital, Beijing, China